CLINICAL TRIAL: NCT04641767
Title: "Fast Heart Fatty Acid Binding Protein (H-FABP) Determination to Rule Out Brain Damage in Mild Traumatic Brain Injury (TBI): the First Multicenter Study Using a Point of Care Device at Trauma and Pediatric Emergency Departments."
Brief Title: BIOmarkers of TRAumatic Brain Injury Spain (BIOTRABIS)
Acronym: BIOTRABIS
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Virgen Macarena (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); Germans Trias i Pujol Hospital (Other); Hospital Sant Joan de Deu (Other); Hospital Universitario La Paz (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Hospital Clinic of Barcelona (Other); Complejo Hospitalario La Mancha Centro (Other); Hospital Son Espases (Other); Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Joan Montaner Villalonga, Joan Montaner, MD, PhD, Hospital Universitario Virgen Macarena
Other Study IDs: BIOTRABIS_FMM-AP171562019
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Mild Traumatic Brain Injury; Moderate Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BIOTRABIS>18 - Pathologic patients: Group that includes adult patients under study. Those with mild TBI will be recruited. In order to determine the severity of the mild TBI, the doctor uses a scale called the Glasgow GCS scale and mild TBI is understood as those with GCS: 14-15.
- BIOTRABIS>18 - Control patients: Group that includes adult control patients. Those with very mild TBI will be recruited (GCS: 15) without symptoms
- BIOTRABIS<18 - Pathologic patients: Group of paediatric patients under study. This will recruit those who come to the emergency department with mild TBI (GCS 14-15) or moderate (GCS 9-13).
- BIOTRABIS<18 - Control patients: Group that includes paediatric control patients. Those with very mild TBI will be recruited (GCS: 15) without symptoms

SUMMARY:
Traumatic brain injury (TBI) is defined as a structural alteration of brain function caused by external causes, where mild traumatic brain injury (mTBI) represents approximately 80% of all TBI, and although its prognosis is relatively good, it represents a significant cost to the system due to the need to perform a cranial computed tomography (CT) scan, a test of high economic value and not without risks such as irradiation, especially important and dangerous in the pediatric age.

The investigators aim to set-up a point of-care (POC) device to validate a biomarker (H-FABP) able to diagnose the presence of brain damage in children and adults with mTBI at trauma and paediatric Emergency Departments using a blood sample, in order to save resources and avoid subjecting patients to a potentially damaging imaging test. But also, to assess whether the incorporation of new biomarkers improves the prediction of brain damage that can be done with H-FABP.

For that, the investigators will recruit a 400 patients' cohort with blood samples using the available POC device for H-FABP biomarker.

ELIGIBILITY:
BIOTRABIS>18 (adult patients)

Inclusion Criteria:

* Patients over 18 years old
* Mild TBI patients the first 24 hours after trauma with GCS of 14-15 points.
* Presence of any of the following symptoms:

  * Loss of consciousness less than 30 minutes, the first 20 minutes after trauma
  * Post-traumatic amnesia less than 24 hours, the first 30 minutes after trauma:
  * Persistent headache
  * Nausea / vomiting
  * Vertigo / dizziness
  * Confusion / disorientation

Exclusion Criteria:

* Recent history (<1 month) of TBI
* Refusal to participate in the study
* Evidence of alcohol or other substance intoxication
* Epilepsy
* Schizophrenia

BIOTRABIS<18 (paediatric patients)

Inclusion Criteria:

* Patients between 0 and 17 years old.
* Mild TBI (GCS 14-15) and moderate TBI (GCS 9-13) patients the first 24 hours after trauma.
* Presence of any of the following symptoms:

  * Loss of consciousness less than 30 minutes, the first 20 minutes after trauma
  * Post-traumatic amnesia less than 24 hours, the first 30 minutes after trauma:
  * Persistent headache
  * Nausea / vomiting
  * Vertigo / dizziness
  * Confusion / disorientation

Exclusion Criteria:

* Recent history (<1 month) of TBI
* Refusal to participate in the study
* Evidence of alcohol or other substance intoxication
* Epilepsy
* Schizophrenia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BIOTRABIS> 18: Group that includes adult patients. Those with mild TBI will be recruited. In order to determine the severity of the TBI, the doctor uses a scale called the Glasgow GCS scale and mild TBI is understood as those with GCS: 14-15.
  BIOTRABIS <18: Group of pediatric patients. This will recruit those who come to the emergency department with mild TBI (GCS 14-15) or moderate (GCS 9-13).
  Each group is subdivided into pathological patients (those under study) or control patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Brain damage diagnostic accuracy | through study completion, an average of 2 years
  Brain damage diagnostic in mild TBI patients during hospital admission [% brain damage versus % non brain damage] will be determined by clinical and neuroimaging criteria (CT) at emergency departments arrivals and compared with diagnostic accuracy of a blood biomarker based test.
Brain damage long term diagnostic accuracy | through study completion, an average of 2 years
  Brain damage diagnostic in mild TBI patients after 3 months [% brain damage long term versus % non brain damage long term ] will be determined by Glasgow Outcome Score (GOSe) through telephone call and compared with previous diagnostic accuracy of a blood biomarker based test.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan Deu Barcelona, Esplugues de Llobregat, Barcelona
  - Complejo Hospitalario La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Virgen del Rocio, Seville, Seville
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Infantil Niño Jesus, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen Macarena, Seville